CLINICAL TRIAL: NCT03851211
Title: Prolaris Enhanced Risk Stratification - an ecONomic and clinicAL Evaluation
Acronym: PERSONAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UR17/104867
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One in 8 men will be diagnosed with prostate cancer during their lifetime. The majority of men diagnosed with prostate cancer have early stage disease, which can be managed in a variety of ways, ranging from monitoring to international treatment. However is it not always clear which treatment option is best.

All men with newly diagnosed localised prostate cancer are assigned a disease risk category (low/intermediate/high risk). This is based on clinical findings and prostate biopsy results, but these factors are limited in their ability to distinguish between aggressive and indolent prostate cancers. The current risk grouping can make it difficult to plan appropriate treatment tailored and personalised to the individual patient.

There is evidence reporting overtreatment of localised prostate cancer in the UK. However, many patients with aggressive disease are wrongly assigned a low risk categorisation and are recommended surveillance when better suited to more interventional treatment.

Myriad Genetics have developed a test, called Prolaris which measures how fast cells in a prostate cancer are dividing to assess its aggressiveness. The Prolaris test is performed on routine prostate biopsy tissue, so patients are not subjected to any additional invasive investigations.

In this study, led by Leeds Teaching Hospitals NHS Trust, the aim is find out if the Prolaris® test score helps patients with newly diagnosed prostate cancer and their clinical team make better informed treatment choices that are tailored to the individual patient.

The aim to achieve a Prolaris risk score for 100 patients and determine the impact it has on treatment decision making. The research team will look at how the test fits into routine clinical practice, investigate the clinician and patient views and understanding on the test report and assess the quality of life of patients in the different risk and treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of prostate cancer
* Able to provide informed written consent
* No contraindication to prostate biopsy
* Newly diagnosed treatment-naive patient with histologically proven localised adenocarcinoma of the prostate
* Low or intermediate D'Amico risk prostate cancer
* Sufficient quantity and quality of tissue remains from biopsy to perform genomic testing
* No contraindication to radical treatment if diagnosed with localised prostate cancer
* Estimated life expectancy >10 years

Exclusion Criteria:

* Men with locally advanced, clinical node positive or metastatic disease
* Patients who lack capacity to consent to study participation
* Non-adenocarcinoma prostate cancer histology

Ages: 18 Years to 100 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men who have a diagnosis of prostate cancer on their prostate biopsy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Prolaris test outcome received via report. | 30-60mins
  Results of the test received.
Treatment counselling | 30-60mins
  Feedback of the results of the prolaris test. Consultant Urologist will see each participant in clinic after receipt of the Prolaris test report. They will explain the results to the patient and the patient will have the opportunity to ask any questions that they may have. The patient will then be able to decide on their treatment option.

CONTACTS AND LOCATIONS:
Locations (1):
- St James's University Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom